CLINICAL TRIAL: NCT05296707
Title: Evaluation of the Possible Effect of Inspiratory Muscle Training on Inflammation Markers and Oxidative Stress in Childhood Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Ozden Gokcek, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/16
Record Dates: First submitted 2022-03-03; First posted 2022-03-25 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Asthma in Children; Children, Adult
Keywords: Childhood Asthma; Inspiratory Muscle Training; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory muscle training group (Experimental): Threshold IMT was given this group. Applied for 7 days 6 weeks.
  Interventions: Other: Inspiratory muscle training; Other: Used routine medicine
- Used routine medicine group (Active Comparator): Followed 6 weeks
  Interventions: Other: Used routine medicine
- Control Group (Active Comparator): Health children
  Interventions: Other: Control group

INTERVENTIONS:
Other: Inspiratory muscle training — The MIP/MEP value of the group that will receive inspiratory muscle training was determined and Threshold IMT training was given with 30%.
  In the training, the subjects were asked to sit in a relaxed position with their upper chest and shoulders relaxed.
  After the nose clip was attached, the children were asked to inhale and exhale by tightly closing the mouthpiece of the instrument with their lips.
  A 30-minute training session was carried out for 6 weeks, with 10-15 repetitive breathing apparatus and 5-10 seconds rest breaks every day.
  Arms: Inspiratory muscle training group
Other: Used routine medicine — After the first evaluation was made, a second evaluation was made after 6 weeks of follow-up.
  Arms: Inspiratory muscle training group; Used routine medicine group
Other: Control group — A healthy child compatible with the age and sex of the patient group was evaluated once.
  Arms: Control Group

SUMMARY:
As inflammation and oxidative stress increase in asthma patients, the severity of symptoms and clinical findings increase. Therefore, this study was planned to evaluate the possible effect of inspiratory muscle training (IMT) on inflammation markers and oxidative stress in childhood asthma.

The study included asthma patient; 35 routine medication, 35 drug therapy and inspiratory muscle training (IMT), and 35 healthy total 105 children aged 8-17 years. Demographic information and hemogram values were recorded. Functional capacity was evaluated with the 6-minute walking test, quality of life PedsQL, respiratory muscle strength oral pressure measuring device, respiratory function test, dyspnea severity with Modified Borg Scale. C-Reactive Protein (CRP), Periostin, Transforming Growth Factor-βeta (TGF-β), Total Antioxidant Status (TAS), Total Oxidant Status (TOS), Oxidative Stress Index (OSI) were analyzed. IMT was given with a Threshold IMT device for 7 days/6 weeks at 30% of maximal inspiratory pressure, and then a second evaluation was made.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with asthma,
* Between the ages of 8-17,
* No asthma attack,
* Cooperating with the study,
* Without cerebral palsy, mental retardation or any other major neurological diagnosis,
* Agreeing to participate in the study,
* Cases whose medication has not been changed for at least three weeks.

Exclusion Criteria:

* Presence of kyphoscoliosis that may affect respiration,
* Having advanced postural alignment problem,
* Having mental problems,
* Having neuromuscular disease,
* Making changes in the medications used in the last three weeks,
* Presence of inflammatory diseases such as juvenile idiopathic arthritis.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker | 6 weeks
  We assessed C reaktive protein from Blood sample
Inflammatory marker | 6 weeks
  We assessed TGF-B from Blood sample
Inflammatory marker | 6 weeks
  We assessed Periostin from Blood sample
Oxidative stress | 6 weeks
  We assessed Total oxidative level.
Oxidative stress | 6 weeks
  We assessed total antioxidative level
Oxidative stress | 6 weeks
  We assessed oxidative status index

SECONDARY OUTCOMES:
Pulmonary function test | 6 weeks
  Pulmonary function test was measured with a portable MiniSpirobank device
Respiratory muscle strength | 6 weeks
  Respiratory muscle strength was measured using a portable (micro RPM brand) electronic mouth pressure measuring device according to ATS/ERS criteria
functional capacity | 6 weeks
  functional capacity was assessed 6 MWT
Quality life | 6 weeks
  Quality life was assessed PedsQl

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Karsıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gokcek O, Yurdalan U, Tugay BU, El C, Dogan S. Evaluation of the possible effect of inspiratory muscle training on inflammation markers and oxidative stress in childhood asthma. Eur J Pediatr. 2023 Aug;182(8):3713-3722. doi: 10.1007/s00431-023-05047-4. Epub 2023 Jun 7. PMID 37285069